CLINICAL TRIAL: NCT05015530
Title: Assessment of Sino-nasal Microbial Communities Changes in Adult Patients With Chronic Rhinosinusitis by 16 rRNA Gene Amplicon Sequencing Before and After 1-month Treatment Duration With Healsea® Chronic: an Exploratory Study
Brief Title: Impact of Symbiofilm On Nasal Microbiota
Acronym: ISONAM
Status: Completed | Type: Observational
Sponsor: Lallemand Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: LPH-2102
Record Dates: First submitted 2021-08-12; First posted 2021-08-20 (Actual); Results first posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2023-03

CONDITIONS: Rhinosinusitis Chronic; Microbiome
Keywords: Rhinosinusitis chronic; Adult; Biofilm; 16S rRNA sequencing; Nasal spray; Microbiome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Middle meatus swabs dedicated to nasal DNA extraction from microbiota
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Test Medical Device: Healsea Chronic nasal spray will be administered twice daily (1 puff, 1-2 sec) in each nostril during 30 days
  Interventions: Device: Healsea® Chronic, hypertonic seawater-based nasal spray supplemented with natural Symbiofilm® extract

INTERVENTIONS:
Device: Healsea® Chronic, hypertonic seawater-based nasal spray supplemented with natural Symbiofilm® extract — Healsea® Chronic nasal spray will be administered twice daily (1 puff, 1-2 sec) in each nostril during 30 days

SUMMARY:
Healsea® chronic is CE marked medical device indicated in adults for the treatment of nasal symptoms of chronic rhinosinusitis. This is an hypertonic seawater-based nasal spray supplemented with natural Symbiofilm® extract (0.2%) isolated from marine bacteria. In vitro, Symbiofilm® inhibits at early stage biofilm formation from bacteria found to be more prevalent and abundant in CRS patients (e.g. Staphylococcus aureus, Pseudomonas aeruginosa). This exploratory study is designed with aim to determine if the antibiofilm properties of Symbiofilm® may modify sino-nasal microbiota, impacting α and/ or β diversities.

DETAILED DESCRIPTION:
Chronic rhinosinusitis (CRS) is an inflammation of the nose and paranasal sinuses and is characterized by two or more symptoms, one of which should be either nasal blockage/obstruction/congestion or nasal discharge (anterior/posterior nasal drip), lasting for 12 weeks or longer. In addition, facial pain or pressure and a reduction in the sense of smell can occur. The condition can occur with or without nasal polyps.

Chronic rhinosinusitis (CRS) is a significant health problem and affects 5-12% of the general population.

The physiopathology of CRS is poorly understood with multiple environmental, host and microbial factors being implicated. Putative pathological factors include changes in the microbiota, imbalance of the local or systemic immune system, allergens, toxins and genetic predisposition.

A dysbiosis mechanism has been proposed as modulating inflammation in diseased sinuses. This hypothesis suggests that externally influenced changes in the nasal microbiome can result in dysbiosis, i.e. a shift from a "normal" or "healthy" microbial community structure and that this shift may be responsible for the initiation or maintenance of CRS. For example, the disruption of the commensal biofilm during a viral upper respiratory tract infection can create a niche for pathogenic species to grow. Despite many contradictory statements in the different studies some common trends emerge. Less diversity in the microbial community rather than an increased overall bacterial load seems to characterize CRS compared to the healthy state with no consensus about specific genera indicative of disease. However, anaerobes and S. aureus are found to be significantly more prevalent and abundant in CRS versus healthy controls. Bacterial biofilm is detected on the sinus mucosa in up to 80% of CRS patients and its presence does not imply that it is causing mucosal inflammation. However, in the context of CRS, there are several possible mechanisms by which biofilms may be pro-inflammatory including the release of planktonic organisms and the release of superantigens, which can cause ciliary dysfunction and inhibition of ciliary clearance. Bacterial biofilms are likely a key modulator of the refractory nature of CRS.

Although clinical evidence from well-designed trials is scarce, European Guidelines for chronic rhinosinusitis recommend daily nasal saline irrigation for reduction of the severity of symptoms of CRS. A recent Cochrane analysis has concluded that daily nasal irrigation with hypertonic saline solution is more effective than placebo to improve patient symptoms. The exact mechanisms by which nasal irrigation works are not known. However, most of the experts agree that it is primarily a mechanical intervention leading to direct cleansing of the nasal mucosa. Nevertheless, the efficacy of such solution remains moderate.

Healsea® Chronic is a CE marked medical device indicated in adults for the treatment of nasal symptoms of chronic rhinosinusitis. This is a seawater-based nasal spray supplemented with a natural Symbiofilm® extract (0.02%) isolated from marine bacteria. The nasal solution is hypertonic (NaCl 2.2%). Symbiofilm® is a marine postbiotic comprising active exopolysaccharides with emulsifying properties and in vitro antibiofilm activity. Antibiofilm properties have been demonstrated with the colorimetric microtiter plate assay. In this model, a significant inhibition of biofilm formation by Staphylococcus aureus and Haemophilus influenzae are observed. Detachment properties from human nasal epithelial cells of Staphylococcus aureus and Pseudomonas aeruginosa has also been demonstrated in vitro, suggesting an inhibition of biofilm formation at early stage in this model. Symbiofilm® has no bacteriostatic nor bactericidal activities.

To date, properly designed studies to evaluate the effect of topical therapies on microbiome are scarce so no definite conclusion can be made. In one study, use of saline irrigation with or without budesonideDCI used was not associated with significantly distinct microbiota composition among either controls or post-operative CRS patients with polyp.

This exploratory study is designed with aim to determine if the antibiofilm properties of Symbiofilm® may modify sino-nasal microbiota, impacting α and/ or β diversities. To this end middle meatus swab specimen will be taken from CRS patients before and after treatment with Healsea® Chronic. Bacteria colonization will be assessed using quantitative PCR and 16S rRNA gene sequencing.

Improvement of nasal symptoms and quality of life will be assessed with the Sino-Nasal Outcome Test score-22 (SNOT-22). Post-market vigilance of Healsea® Chronic and vigilance of study procedures will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 - 70 years
2. Provision of signed and dated informed consent form
3. Stated willingness to comply with all study procedures and availability for the duration of the study
4. Diagnosed with CRS based on the diagnostic criteria of the EPOS guideline
5. Registered with a social security scheme or covered by such a regime

Exclusion Criteria:

1. Antibiotics or oral corticosteroids intake in the month prior to the study
2. Endoscopic sinus surgery in the past 6 months
3. Cystic fibrosis
4. Wegener's granulomatosis
5. Immunodeficiency
6. Defective access to middle meatus
7. Lidocaine allergy
8. Known hypersensitivity/allergy to any component of the test device
9. Pregnant/Lactating female or absence of efficient contraception
10. Under tutorship or guardianship

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects will be recruited by the site among outpatients coming for routine consultation because of CRS.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pr Guillaume de Bonnecaze, MD, PhD, Principal Investigator — Department of Otorhinolaryngology , University Hospital of Toulouse (Larrey), France
Locations (1):
- Larrey Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fokkens WJ, Lund VJ, Hopkins C, Hellings PW, Kern R, Reitsma S, Toppila-Salmi S, Bernal-Sprekelsen M, Mullol J, Alobid I, Terezinha Anselmo-Lima W, Bachert C, Baroody F, von Buchwald C, Cervin A, Cohen N, Constantinidis J, De Gabory L, Desrosiers M, Diamant Z, Douglas RG, Gevaert PH, Hafner A, Harvey RJ, Joos GF, Kalogjera L, Knill A, Kocks JH, Landis BN, Limpens J, Lebeer S, Lourenco O, Meco C, Matricardi PM, O'Mahony L, Philpott CM, Ryan D, Schlosser R, Senior B, Smith TL, Teeling T, Tomazic PV, Wang DY, Wang D, Zhang L, Agius AM, Ahlstrom-Emanuelsson C, Alabri R, Albu S, Alhabash S, Aleksic A, Aloulah M, Al-Qudah M, Alsaleh S, Baban MA, Baudoin T, Balvers T, Battaglia P, Bedoya JD, Beule A, Bofares KM, Braverman I, Brozek-Madry E, Richard B, Callejas C, Carrie S, Caulley L, Chussi D, de Corso E, Coste A, El Hadi U, Elfarouk A, Eloy PH, Farrokhi S, Felisati G, Ferrari MD, Fishchuk R, Grayson W, Goncalves PM, Grdinic B, Grgic V, Hamizan AW, Heinichen JV, Husain S, Ping TI, Ivaska J, Jakimovska F, Jovancevic L, Kakande E, Kamel R, Karpischenko S, Kariyawasam HH, Kawauchi H, Kjeldsen A, Klimek L, Krzeski A, Kopacheva Barsova G, Kim SW, Lal D, Letort JJ, Lopatin A, Mahdjoubi A, Mesbahi A, Netkovski J, Nyenbue Tshipukane D, Obando-Valverde A, Okano M, Onerci M, Ong YK, Orlandi R, Otori N, Ouennoughy K, Ozkan M, Peric A, Plzak J, Prokopakis E, Prepageran N, Psaltis A, Pugin B, Raftopulos M, Rombaux P, Riechelmann H, Sahtout S, Sarafoleanu CC, Searyoh K, Rhee CS, Shi J, Shkoukani M, Shukuryan AK, Sicak M, Smyth D, Sindvongs K, Soklic Kosak T, Stjarne P, Sutikno B, Steinsvag S, Tantilipikorn P, Thanaviratananich S, Tran T, Urbancic J, Valiulius A, Vasquez de Aparicio C, Vicheva D, Virkkula PM, Vicente G, Voegels R, Wagenmann MM, Wardani RS, Welge-Lussen A, Witterick I, Wright E, Zabolotniy D, Zsolt B, Zwetsloot CP. European Position Paper on Rhinosinusitis and Nasal Polyps 2020. Rhinology. 2020 Feb 20;58(Suppl S29):1-464. doi: 10.4193/Rhin20.600. PMID 32077450
- [Background] Sivasubramaniam R, Douglas R. The microbiome and chronic rhinosinusitis. World J Otorhinolaryngol Head Neck Surg. 2018 Oct 31;4(3):216-221. doi: 10.1016/j.wjorl.2018.08.004. eCollection 2018 Sep. PMID 30506054
- [Background] Boase S, Foreman A, Cleland E, Tan L, Melton-Kreft R, Pant H, Hu FZ, Ehrlich GD, Wormald PJ. The microbiome of chronic rhinosinusitis: culture, molecular diagnostics and biofilm detection. BMC Infect Dis. 2013 May 8;13:210. doi: 10.1186/1471-2334-13-210. PMID 23656607
- [Background] Ramakrishnan VR, Hauser LJ, Frank DN. The sinonasal bacterial microbiome in health and disease. Curr Opin Otolaryngol Head Neck Surg. 2016 Feb;24(1):20-5. doi: 10.1097/MOO.0000000000000221. PMID 26575518
- [Background] Hoggard M, Wagner Mackenzie B, Jain R, Taylor MW, Biswas K, Douglas RG. Chronic Rhinosinusitis and the Evolving Understanding of Microbial Ecology in Chronic Inflammatory Mucosal Disease. Clin Microbiol Rev. 2017 Jan;30(1):321-348. doi: 10.1128/CMR.00060-16. PMID 27903594
- [Background] Koeller K, Herlemann DPR, Schuldt T, Ovari A, Guder E, Podbielski A, Kreikemeyer B, Olzowy B. Microbiome and Culture Based Analysis of Chronic Rhinosinusitis Compared to Healthy Sinus Mucosa. Front Microbiol. 2018 Apr 17;9:643. doi: 10.3389/fmicb.2018.00643. eCollection 2018. PMID 29755418
- [Background] Fastenberg JH, Hsueh WD, Mustafa A, Akbar NA, Abuzeid WM. Biofilms in chronic rhinosinusitis: Pathophysiology and therapeutic strategies. World J Otorhinolaryngol Head Neck Surg. 2016 May 5;2(4):219-229. doi: 10.1016/j.wjorl.2016.03.002. eCollection 2016 Dec. PMID 29204570
- [Background] Chong LY, Head K, Hopkins C, Philpott C, Glew S, Scadding G, Burton MJ, Schilder AG. Saline irrigation for chronic rhinosinusitis. Cochrane Database Syst Rev. 2016 Apr 26;4(4):CD011995. doi: 10.1002/14651858.CD011995.pub2. PMID 27115216
- [Background] O'Toole GA. Microtiter dish biofilm formation assay. J Vis Exp. 2011 Jan 30;(47):2437. doi: 10.3791/2437. PMID 21307833
- [Background] Liu CM, Kohanski MA, Mendiola M, Soldanova K, Dwan MG, Lester R, Nordstrom L, Price LB, Lane AP. Impact of saline irrigation and topical corticosteroids on the postsurgical sinonasal microbiota. Int Forum Allergy Rhinol. 2015 Mar;5(3):185-90. doi: 10.1002/alr.21467. Epub 2014 Dec 29. PMID 25556553
- [Background] Hopkins C, Gillett S, Slack R, Lund VJ, Browne JP. Psychometric validity of the 22-item Sinonasal Outcome Test. Clin Otolaryngol. 2009 Oct;34(5):447-54. doi: 10.1111/j.1749-4486.2009.01995.x. PMID 19793277

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subjects will be recruited by the site among outpatients coming for routine consultation because of CRS. The first patient was screened and enrolled on 12th December 2022, the last patient was screened and enrolled on 25th April 2023.
Groups:
- Healsea® Chronic: Hypertonic Seawater-Based Nasal Spray With Natural Symbiofilm® Extract: Healsea® Chronic nasal spray will be administered twice a day (1 puff, 1-2 sec) in each nostril during 30 days.
Period: Overall Study
Arm/Group | Healsea® Chronic: Hypertonic Seawater-Based Nasal Spray With Natural Symbiofilm® Extract
Started | 12
Safety Set (All subjects who will have used the investigational medical device at least once.) | 12
Full Analysis Set (FAS) (All subjects from the Safety Set who will have at least one post baseline Sino Nasal Outcome Test-22 (SNOT-22) evaluation.) | 12
Per Protocol Set (PP) (All subjects from the FAS without any major protocol deviation.) | 3
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healsea® Chronic: Hypertonic Seawater-Based Nasal Spray With Natural Symbiofilm® Extract
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 12
Region of Enrollment [Number; unit: participants]
  France | 12
Baseline SNOT-22 (total) [Mean (Standard Deviation); unit: score on a scale] — The SNOT-22 is a validated patient-reported outcome measure that captures the physical, functional,and emotional consequences of rhinosinusitis. Patients should rate sino-nasal symptoms and their impact from 0 to 5 where 0 means that there is no complaint and 5 means that there are serious complaints. The SNOT-22 score is calculated as the sum of scores provided for each question and ranges from 0 (no complaint at all) to 110.
  score on a scale | 59.3 (21.2)
α diversity [Mean (Standard Deviation); unit: Shannon Index] — The alpha diversity is a quantitative index measure that reflects the diversity of bacterial species in a sample. The diversity of microbiota present in the given sample was measured using the Shannon index. The greater Shannon index value, the more diverse nasal microbiota.
  Shannon Index | 2.041 (0.900)

OUTCOME MEASURES:

1. Primary Outcome: Comparaison of Alpha-diversity of Sino-nasal Microbiota Before and After Treatment (Visit 1 and Visit 2)
Description: Comparaison of the values of alpha diversity of bacterial species assessed by the Shannon index at baseline and after the treatment period
Time Frame: At baseline (V1) and at end of the 30-day treatment period (V2)
Population: Full Analysis Population
Measure: Mean (Standard Deviation); unit: Shannon Index
Groups:
- Healsea® Chronic Baseline Value: Shannon index before administration of Healsea® Chronic
- Healsea® Chronic After 30-day Treatment: Shannon index after administration of Healsea® Chronic twice a day (1 puff, 1-2 sec) in each nostril during 30 days.
Arm/Group | Healsea® Chronic Baseline Value | Healsea® Chronic After 30-day Treatment
Number analyzed (Participants) | 12 | 12
Shannon Index | 2.041 (0.900) | 2.114 (1.041)
Statistical Analysis 1: Comparison: Healsea® Chronic Baseline Value vs Healsea® Chronic After 30-day Treatment; α-diversity assessed using the Kruskal-Wallis test; Test type: Superiority; p = 0.908, Kruskal-Wallis

2. Secondary Outcome: Impact of Healsea® Chronic on Quality of Life Assessed by the Sino-Nasal Outcome Test Score-22
Description: Change of SNOT-22 total score at the end of the 30-day treatment period versus baseline . A change >-9 is deemed clinically meaningful.
Time Frame: End of treatment (Visit 2(V2)-Day 30) versus screening/inclusion (Visit 1(V1)-Day 1)
Population: Full Analysis Population
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Healsea Chronic Nasal Spray Baseline Value: Value of SNOT-22 before administration of Healsea Chronic
- Healsea® Chronic Nasal Spray After 30 Days: SNOT-22 total score after administration of Healsea® Chronic twice a day (1 puff, 1-2 sec) in each nostril during 30 days.
Arm/Group | Healsea Chronic Nasal Spray Baseline Value | Healsea® Chronic Nasal Spray After 30 Days
Number analyzed (Participants) | 12 | 12
score on a scale
  Absolute values of SNOT-22 total score | 59.3 (21.2) | 41.8 (25.5)
  Change of SNOT-22 total score versus baseline | 0 (0) | -17.5 (17)

3. Secondary Outcome: Patient Satisfaction Questionnaire (Usability)
Description: To assess patient 's satisfaction regarding the medical device usability
Time Frame: Visit 2(V2)-Day 30 (end of treatment)
Population: Full Analysis Population
Measure: Count of Participants; unit: Participants
Arm/Group | Healsea® Chronic: Hypertonic Seawater-Based Nasal Spray With Natural Symbiofilm® Extract
Number analyzed (Participants) | 12
Participants
  Missing | 0
  Not easy | 0
  Pretty easy | 0
  Easy | 0
  Very easy | 12

4. Secondary Outcome: Patient Satisfaction Questionnaire (Taste)
Description: To assess patient 's satisfaction regarding the sensory perception (residual taste after spraying)
Time Frame: Visit 2(V2)-Day 30 (end of treatment)
Population: Full Analysis Population
Measure: Count of Participants; unit: Participants
Arm/Group | Healsea® Chronic: Hypertonic Seawater-Based Nasal Spray With Natural Symbiofilm® Extract
Number analyzed (Participants) | 12
Participants
  Missing | 0
  Not pleasant | 0
  Neutral | 8
  Pleasant | 3
  Very pleasant | 1

5. Secondary Outcome: Patient Satisfaction Questionnaire (Efficacy)
Description: To assess patient 's satisfaction regarding product efficacy for chronic Rhinosinusitis (Cleansing and Moistening of nasal mucosa)
Time Frame: Visit 2(V2)-Day 30 (end of treatment)
Population: Full Analysis Population
Measure: Count of Participants; unit: Participants
Arm/Group | Healsea® Chronic: Hypertonic Seawater-Based Nasal Spray With Natural Symbiofilm® Extract
Number analyzed (Participants) | 12
Participants
  Missing | 0
  No improvement | 0
  Slight improvement | 2
  Moderate improvement | 6
  Very clear improvement | 4

6. Other Pre Specified Outcome: Reporting of Adverse Events, Incidents and Expected Side Effects
Description: Assessment of materiovigilance from the medical device (incidents, expected side effects) and reporting of adverse reactions related to the additional invasive procedure (swab of the nasal meatus)
Time Frame: During the intervention, up to 30 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events/incidents were collected during the intervention and up to 30 days
Description: In this investigation with a medical device, 3 types of adverse events were to be reported: non-related/related adverse events and serious adverse events related to the invasive procedure. No SAE has been reported.
  Also, materiovigilance from the medical device (incidents, expected side effects) was to be reported. One incident was reported: Headache (Nervous system disorders).
Arm/Group | Healsea® Chronic: Hypertonic Seawater-Based Nasal Spray With Natural Symbiofilm® Extract
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healsea® Chronic: Hypertonic Seawater-Based Nasal Spray With Natural Symbiofilm® Extract (N=12)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Palatal disorder (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Small number of subjects (12 VS 20 expected)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/30/NCT05015530/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-04): https://cdn.clinicaltrials.gov/large-docs/30/NCT05015530/SAP_001.pdf